CLINICAL TRIAL: NCT00623753
Title: Evaluate Tolerability and Safety of Multi-Envelope, Prime-boost HIV Vaccine (DVP) in Healthy Adults
Brief Title: Evaluate Tolerability of a Multi-envelope, Prime-boost HIV Vaccine in Healthy Adults
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DVP-I
Record Dates: First submitted 2008-02-18; First posted 2008-02-26 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2011-09

CONDITIONS: HIV Infections
Keywords: Vaccine; Prevention; HIV; AIDS; Human Immunodeficiency Virus; HIV Seronegativity, HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Biological: EnvDNA, PolyEnv1, EnvPro

INTERVENTIONS:
Biological: EnvDNA, PolyEnv1, EnvPro — Description: The vaccine regimen is a series of 6 injections given 28 days apart. EnvDNA is administered intramuscularly as 100 mcg of recombinant DNA in 1.5 mL of PBS as injections #1, 2 and 5. PolyEnv1 is recombinant vaccinia virus administered subcutaneously as 107 pfu in 0.8 mL of PBS as injection #3. EnvPro is administered intramuscularly as 100 mcg of recombinant protein and 500 mcg of aluminum hydroxide (alum) adjuvant in 1.0 mL of PBS as injections #4 and 6.

SUMMARY:
Vaccines have been very successful in preventing viral infections such as hepatitis B and the measles. Viral vaccines work by causing a person's immune system to make cells that will work against the virus. Due to the success in treating other viral infections, scientists are trying to develop a vaccine for human immunodeficiency virus (HIV). HIV infection is the cause of acquired immune deficiency syndrome (AIDS). AIDS is one of the most serious viral infections we know.

This is a research study to evaluate the safety of a possible vaccine against HIV. Researchers want to determine that a person's immune system can respond to the HIV before he or she is exposed to it. Therefore that person may be able to be protected from infection with HIV.

DETAILED DESCRIPTION:
This is a research study to find out about the safety of a new potential vaccine regimen against HIV. This potential vaccine regimen consists of a sequence of six vaccine shots that are being studied to see if they can help to protect people from the human immunodeficiency virus (HIV). HIV infection is the cause of AIDS. AIDS is one of the most serious viral infections we know. Twenty million people around the world have already died of AIDS and over 40 million people are currently infected with the virus. This study is being done to help us find an HIV vaccine that works.

Vaccines have been very successful in preventing other viral infections, such as hepatitis B, polio, and measles. Viral vaccines work by causing a person's immune system to make antibodies and immune cells against the virus or to "respond" to the virus. Because of the success with other viral infections, scientists are trying to develop a successful vaccine for HIV. If a person's immune system can respond to HIV before he or she is exposed to it, that person may be able to be protected from infection with HIV.

The vaccine regimen that will be tested in this study is based on the information that the virus uses to make a small part of the HIV. This small part is called the "envelope" or coating around the virus. Because only the information for this one part of the virus is used in the vaccine, the vaccine cannot cause HIV infection. We make all parts of the vaccine regimen in test tubes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults; age > 18 years, born after 1972 if born in U.S.
* Informed consent
* Normal history and physical exam
* HIV-1 negative as documented by ELISA and Western blot analysis within 30 days prior to immunization
* Normal laboratory values within 60 days prior to immunization defined as:

  * hemoglobin greater than or equal to 12.0 gm/dl for females and greater than or equal to 14.0 gm/dl for males
  * White blood cell count > 3500 cells/mm3
  * Platelet count 150,000 - 550,000 cells/mm3
  * Absolute CD4+ count > 400 cells/mm3
  * AST and ALT within normal institutional limits
  * Serum creatinine within normal institutional limits
* Normal CPK-MB (creatine kinase isoenzyme MB) and troponin I within 30 days prior to immunization
* Normal ECG within 30 days prior to immunization
* No evidence of smallpox vaccination (born in the U.S. after 1972 with no typical scar on the deltoid, ankle, thigh or between the scapulae and no history of vaccination in personal immunization record)
* No entry into military service before 1990
* Fewer than 3 of the following:

  * Current cigarette smoker
  * History of high cholesterol
  * History of diabetes or high blood sugar
  * High blood pressure
  * Heart disease before age 50 in parent or sibling
* Not planning to become pregnant during study vaccinations and for 3 months after last vaccination
* Vaccinia virus seronegative

Exclusion Criteria:

* History of immunosuppressive illness, chronic illness (e.g. asthma, bleeding diathesis, etc) or use of any immunosuppressive medications (e.g. steroids)
* History of neurological disorder
* Receiving therapy or prophylaxis for tuberculosis
* Known allergy to the antibiotic kanamycin
* History of eczema, atopic dermatitis and other acute, chronic or exfoliative conditions
* Household contact with persons with eczema or other exfoliative skin conditions
* Pregnant or nursing women
* Household contact with persons with immunodeficiency (including eczema or use of immunosuppressive medications)
* Household contact with persons less than 12 months of age
* Household contact with pregnant women
* History of cardiac disease such as previous myocardial infarction, angina, congestive heart failure, or cardiomyopathy
* Any member of the Investigator's laboratory program
* Participation in previous HIV vaccine trial

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2007-05; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the tolerability and safety of the multi-envelope vaccine regimen. | 1 year

SECONDARY OUTCOMES:
To characterize the kinetics, duration and magnitude of the HIV-envelope specific immune responses elicited by the multi-envelope vaccine regimen. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pat Flynn, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org